CLINICAL TRIAL: NCT05689645
Title: F573 for Injection for the Treatment of Liver Injury/Failure : Randomized, Double-blind, Placebo-controlled Phase Ⅱa Clinical Trial
Brief Title: F573 for Injection for the Treatment of Liver Injury/Failure
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KDN-F573-202202
Record Dates: First submitted 2022-12-05; First posted 2023-01-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Acute Liver Failure; Acute-On-Chronic Liver Failure
Keywords: F573 for injection Liver Injury/Failure
MeSH Terms: conditions — Liver Failure, Acute; Acute-On-Chronic Liver Failure | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F573 for injection groups (Experimental): The first stage:the first 16 patients with liver injury were given doses of 0.5, 1.0 and 2.0 mg/kg, and the subsequent 9 patients with CHB were given doses of 2.0 mg/kg, with an administration volume of 2 mL and intramuscular injection (IM) according to the efficacy and safety test results of the first 16 patients. The dose was given once a day for 7 days and calculated according to the weight of the last visit.
  The second stage:According to the results of Phase I efficacy and safety trials, the dosage was determined to be 0.5 mg/kg and 2.0 mg/kg, the dosage volume was 2 mL, intramuscular injection (IM), once a day for 14 days, and the dosage was calculated according to the weight of the latest visit.
  The third stage:The dosage was determined according to the results of the first and second phase efficacy and safety trials. The dosage volume was 2 mL, intramuscular injection (IM), once a day for 28 consecutive days, and the dosage was calculated according to the weight of the latest
  Interventions: Drug: F573 for injection
- Placebo Comparator (Placebo Comparator): 1. The first stage: The dosage was 2 mL by intramuscular injection (IM) once a day for 7 days.
     Basic treatment: enteric-coated diammonium glycyrrhizinate capsules were administered at a dose of 150 mg 3 times a day.
  2. The second stage: The dosage was 2 mL by intramuscular injection (IM) once a day for 14 days.
     Basic treatment: Polyene phosphatidylcholines and glutathione drugs (no restricted dosage forms) are accepted as basic treatment.
  3. The third stage: the Screen eligible subjects were treated with Sterilizing water for injection. The dose volume was 2 mL, intramuscular injection (IM), once a day for 28 consecutive days. Basic treatment: receive acetylcysteine injection at a dose of 8 g / d once a day.
  Interventions: Drug: Sterilizing water for injection

INTERVENTIONS:
Drug: F573 for injection — The first stage:the first 16 patients with liver injury were given doses of 0.5, 1.0 and 2.0 mg/kg, and the subsequent 9 patients with CHB were given doses of 2.0 mg/kg, with an administration volume of 2 mL and intramuscular injection (IM) according to the efficacy and safety test results of the first 16 patients. The dose was given once a day for 7 days and calculated according to the weight of the last visit.
  The second stage:According to the results of Phase I efficacy and safety trials, the dosage was determined to be 0.5 mg/kg and 2.0 mg/kg, the dosage volume was 2 mL, intramuscular injection (IM), once a day for 14 days, and the dosage was calculated according to the weight of the latest visit.
  The third stage:The dosage was determined according to the results of the first and second phase efficacy and safety trials. The dosage volume was 2 mL, intramuscular injection (IM), once a day for 28 consecutive days, and the dosage was calculated according to the weight of the latest .
  Arms: F573 for injection groups
Drug: Sterilizing water for injection — The composition of this product is water for injection, and the dosage volume is 2mL for intramuscular injection.
  Medication course: The first stages were administered once a day for 7 days and second stages were administered once a day for 14 days. The third stage was administered once a day for 28 days.
  Arms: Placebo Comparator

SUMMARY:
This study was a randomized, double-blind, placebo-controlled PhaseⅡ clinical trial .

The primary objective of this study was to evaluate the safety of F573 for injection in patients with liver injury (drug-induced liver injury (DILI), chronic hepatitis B (CHB), intrahepatic cholestatic liver injury, etc.).

DETAILED DESCRIPTION:
In a randomized, double-blind, placebo-controlled design, the study was divided into two phases according to the subjects' risk of liver failure due to liver injury.

The first stage: Twenty-five patients with liver injury (DILI patients and other types of patients with the same degree of liver injury) were enrolled. The trial was first conducted in 16 participants who were treated with the experimental drug or placebo at a 1:1:1:1 ratio of 0.5, 1.0, and 2.0 mg/kg. Then, 9 patients with CHB were treated with the experimental drug, and the dose was determined to be 2.0 mg/kg according to the efficacy and safety test results of the 16 patients enrolled first.After subject consent is obtained, pharmacokinetic blood samples will be collected from 9 CHB patients subsequently enrolled in Phase I.

The second stage:A total of 24 patients with liver injury (DILI patients and intrahepatic cholestasis type liver injury) were enrolled, and qualified subjects were treated with the experimental drug or placebo in a ratio of 3:1, once a day for 14 days. The dosage was determined to be 0.5 mg/kg and 2.0 mg/kg based on the results of phase I efficacy and safety trials. First, a trial was conducted in the 0.5 mg/kg dose group, and 12 subjects were enrolled and treated with the test drug or placebo at a ratio of 3:1, once a day for 14 days. After the 0.5 mg/kg dose group was completed, the experiment of 2.0 mg/kg dose group was carried out. 12 subjects were also enrolled and received the test drug or placebo in a ratio of 3:1, once a day for 14 days.

The Third stage:

The study was randomized, double-blind, placebo-controlled. The study was divided into a screening period (14 days), treatment period (28 days), and follow-up period (90 days).

Eligible subjects were given the experimental drug or placebo in a ratio of 3:1, once a day for 28 days, and the dose was determined according to the efficacy and safety results of phase I and Phase II trials. Subjects also received the drug acetyl cysteine injection (NAC). After discontinuation, participants were followed for 90 days for safety. During the study, subjects were visited at planned sites for clinical laboratory examination, vital signs, physical examination, 12-lead electrocardiography, abdominal B-ultrasonography, cardiac color ultrasonography, biomarker testing, MELD score, AARC score, survival status assessment, monitoring of AE, and recording of subjects' concomitant/concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

（1）The first stage:

Participants who meet all of the following criteria will be enrolled in the study:

1. Age ≥18 and ≤60 years old, gender is not limited;
2. Patients with liver injury clinically diagnosed with hepatocyte injury or mixed liver injury or CHB patients with hepatitis B virus infection for more than 6 months (refer to the "Chronic Hepatitis B Prevention and Treatment Guidelines (2019 edition)"). Screening patients with CHB may provide etiological (HBsAg positive and/or HBV DNA positive) or clinical or pathological evidence (liver tissue biopsy results) that HBV infection has been present for more than 6 months.
3. Serum ALT: 2~ 10× upper limit of normal (ULN), TBil: <5×ULN;
4. DILI patients: the abnormal duration of liver biochemical indexes [ALT, AST, ALP, gamma-glutamyltranspeptides (GGT), TBil, albumin, prothrombin time] does not exceed 90 days;
5. The subject (including the partner) is willing to take effective contraceptive measures from the screening until 6 months after the last test drug administration;
6. Sign informed consent and be able to comply with the requirements of the program; If the subject is unable to sign the informed consent form, it must be signed by a legal guardian or witness as required by the regulations.

(2)The second stage:

Subjects meeting all of the following criteria will be included in the study:

1. Age ≥ 18 and ≤ 65 years old, with no gender restrictions;
2. According to the "Chinese Guidelines for the Diagnosis and Treatment of Drug-Induced Liver Injury (2023 Edition)", patients diagnosed with drug-induced liver injury (DILI) or those diagnosed with intrahepatic cholestasis type liver injury. Patients with DILI and intrahepatic cholestasis type liver injury need to meet the following criteria separately;

   1. Patients with DILI need to simultaneously meet the following conditions: ① Serum ALT > 3 times the upper limit of normal (ULN), and TBil > 2 times the ULN (the ULN of TBil refers to 17.1 μmol/L according to international standards); ② Abnormal liver biochemical indicators (ALT, AST, ALP, TBil) persist for no more than 60 days;
   2. Patients with intrahepatic cholestasis type liver injury need to simultaneously meet the following conditions: ① TBil > 2 times the ULN (the ULN of TBil refers to 17.1 μmol/L); ② ALP > 1.5 times the ULN; ③ALT>1×ULN;
3. The subjects (including their partners) are willing to voluntarily adopt effective contraceptive measures from the time of the initial screening until 6 months after the last administration of the investigational drug;
4. They have signed the informed consent form and can comply with the requirements of the protocol; if the subjects are unable to sign the informed consent form, it must be signed by a legal guardian or a witness as required by the regulations.

The third stage:

Subjects who meet all of the following criteria will be enrolled in the study:

1. Age ≥18 and ≤70 years old, gender is not limited; 2. Patients diagnosed with chronic and acute liver failure with TBil≥5×ULN according to the "Guidelines for Diagnosis and Treatment of Liver Failure (2018 Edition)" may have hepatic encephalopathy (Grade 1-2) or ascites (grade 1-2) 4 weeks before subject screening. And 5≤AARC score ≤10 (AARC rating I-II); 3. The subject (including the partner) is willing to take effective contraceptive measures from the screening until 6 months after the last trial drug administration; 4. Sign informed consent and comply with the requirements of the program; If the subject is unable to sign the informed consent form, it must be signed by a legal guardian or witness as required by the regulations.

-

Exclusion Criteria:

The first stage:

Subjects meeting one of the following conditions will not be included in the trial:

1. According to the investigator's judgment, the subjects were patients with cholestatic liver injury;
2. Previous diagnosis of cirrhosis or liver hardness determination (LSM) at screening ≥ 12.4kPa;
3. Patients with severe or life-threatening heart, lung, brain, kidney, gastrointestinal and systemic diseases, and patients with malignant tumors;
4. There are the following laboratory test values or abnormal test values:

   1. Blood routine: platelet (PLT) <75× 109/L, hemoglobin (HGB) <90 g/L;
   2. Prothrombin activity <40%, prothrombin time (PT) extended >5 s;
   3. Left ventricular ejection fraction (LVEF) <50%;
5. Allergic or intolerant to the investigational drug, or allergic;
6. The subject is unable to express his main complaint, such as mental illness and severe neurosis;
7. Poor compliance can not partner;
8. Pregnant women, breastfeeding women or women of childbearing age who are trying to conceive;
9. Participants in other clinical trials within 3 months;
10. Patients who had used liver protection drugs other than ursodeoxycholic acid or adenosylmethionine within 3 days before randomization;
11. The researcher considers any circumstances unsuitable for inclusion.

The second stage:

Subjects meeting one of the following conditions will not be included in the trial:

1. The diagnosis is advanced liver cirrhosis (with complications such as ascites and hepatic encephalopathy), or liver cancer, or when liver stiffness measurement (LSM) is ≥ 18.0 kPa during screening.
2. Patients with severe or life-threatening heart, lung, brain, kidney, gastrointestinal and systemic diseases are malignantTumor patients;
3. There are the following laboratory test values or abnormal test values:

   1. Blood routine: platelet (PLT) <100×109/L, hemoglobin (HGB) <100 g/L;
   2. INR>1.4, or as determined by the investigator to meet the criteria for severe hepatitis;
   3. Left ventricular ejection fraction (LVEF) <50%;
4. Allergic or intolerant to the investigational drug, or allergic;
5. The subject is unable to express his main complaint, such as mental illness and severe neurosis;
6. Poor compliance can not partner;
7. Pregnant women, breastfeeding women or women of childbearing age who are trying to conceive;
8. Participants in other clinical trials within 3 months;
9. Patients who had used liver protection drugs other than ursodeoxycholic acid or adenosylmethionine and basic therapeutic drugs (polyene phosphatidylcholines and glutathione drugs) within 3 days before randomization;
10. Patients who had used glucocorticoids or interferon drugs within 3 days before randomization;
11. The researcher considers any circumstances unsuitable for inclusion.

The third stage:

Subjects meeting one of the following conditions will not be included in the trial:

1. Patients who have completed liver transplantation or plan to undergo liver transplantation within 1 month;
2. Severe grade 3 ascites or stubborn ascites;
3. Patients with ≥ grade 3 hepatic encephalopathy;
4. Patients who received artificial liver treatment within 1 week before screening;
5. Patients with severe underlying diseases, such as respiratory system, digestive system, circulatory system, endocrine and other diseases and malignant tumors, and patients with severe infections that cannot be controlled by drugs;
6. During the screening period or within 1 month before screening, the results of gastroscopy or imaging (abdominal B-ultrasound, CT or MRI) examination suggest severe varicose veins with bleeding risk;
7. Patients with acute kidney injury (AKI), defined as meeting one of the following conditions:

   1. Serum creatinine (Scr) increased ≥26.5 μmol/L (0.3 mg/dL, 1 mg/dL=88.4 μmol/L) within 48 h;
   2. The Scr increase exceeds 1.5 times or more of the base value within 7 days;
   3. Decreased urine volume (<0.5 mL/kg/h) for more than 6 hours;
8. Allergic or intolerant to the investigational drug, or allergic;
9. The subject is unable to express his main complaint, such as mental illness and severe neurosis;
10. Poor compliance can not partner; 11 Pregnant women, breastfeeding women or women of childbearing age who are trying to conceive;

12. Participants in other clinical trials within 3 months; 13. The researcher considers any circumstances unsuitable for inclusion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE), serious adverse events (SAE) | 7 days of administration in the first stage and 14 days of administration in the second stage
  to record Adverse events and serious adverse events in the trial
Adverse events (AE), serious adverse events (SAE) | followed up for 28 days in the first stage and followed up for 14 days in the second stage
  to record Adverse events and serious adverse events in the trial
clinical laboratory tests ：blood routine | 7 days of administration in the first stage and 14 days of administration in the second stage
  blood routine report contains the following values: RBC,WBC,NE%,LY%,HGB,PLT.
clinical laboratory tests ：blood routine | followed up for 28 days in the first stage and followed up for 14 days in the second stage
  blood routine report contains the following values: RBC,WBC,NE%,LY%,HGB,PLT.
clinical laboratory tests ：blood biochemistry | 7 days of administration in the first stage and 14 days of administration in the second stage
  blood biochemistry report contains the following values: DBIL,TBIL,Urea，BUN,Cr，AST，ALT，GGT, TP, ALB, GLU,TG, TC, K,Na,CI, UA,LDH, ALP, PAB, RBP, AFP.
clinical laboratory tests ：blood biochemistry | followed up for 28 days in the first stage and followed up for 14 days in the second stage
  blood biochemistry report contains the following values: DBIL,TBIL,Urea，BUN,Cr，AST，ALT，GGT, TP, ALB, GLU,TG, TC, K,Na,CI, UA,LDH, ALP, PAB, RBP, AFP.
clinical laboratory tests : urine routine | 7 days of administration in the first stage and 14 days of administration in the second stage
  urine routine report contains the following values: GLU,PRO,RBC,WBC.
clinical laboratory tests : urine routine | followed up for 28 days in the first stage and followed up for 14 days in the second stage
  urine routine report contains the following values: GLU,PRO,RBC,WBC.
clinical laboratory tests ：blood coagulation function | 7 days of administration in the first stage and 14 days of administration in the second stage
  blood coagulation function report contains the following values: TT, APTT, PT, INR.
clinical laboratory tests ：blood coagulation function | followed up for 28 days in the first stage and followed up for 14 days in the second stage
  blood coagulation function report contains the following values: TT, APTT, PT, INR.
12-lead electrocardiogram (ECG) | 7 days of administration in the first stage and 14 days of administration in the second stage
  12-lead electrocardiogram (ECG) report contains the following values: HR, BP,DP,PR intervals,QRS intervals,QT intervals,QTc intervals.
12-lead electrocardiogram (ECG) | followed up for 28 days in the first stage and followed up for 14 days in the second stage
  12-lead electrocardiogram (ECG) report contains the following values: HR, BP,DP,PR intervals,QRS intervals,QT intervals,QTc intervals.
All-cause mortality | 28 days after completion of dosing in the third stage
  All-cause mortality within 28 days after completion of dosing.
All-cause mortality | 90 days after completion of dosing in the third stage
  All-cause mortality within 90 days after completion of dosing.

SECONDARY OUTCOMES:
Basin alanine aminotransferase (ALT) | after 7 days of administration in the first and second stages
  ALT values reflect hepatocyte injury
Basin alanine aminotransferase (ALT) | after 14 days of administration in the second stages
  ALT values reflect hepatocyte injury
Basin alanine aminotransferase (ALT) | followed up for 28 days in the first stage and followed up for 14 days in the second stage
  ALT values reflect hepatocyte injury
peak concentration (Cmax) | 12 hours after administration in the first and second stages
  Pharmacokinetic parameters: peak concentration (Cmax).
Peak-reaching time (Tmax) | 12 hours after administration in the first and second stages
  Pharmacokinetic parameters: Peak-reaching time (Tmax)
half-life period (T1/2) | 12 hours after administration in the first and second stages
  Pharmacokinetic parameters: half-life period (T1/2)
Blood concentration-area (AUC) | 12 hours after administration in the first and second stages
  Blood concentration-area (AUC) under the time curve from zero to t0-t), Area under the blood concentration-time curve from 0 to infinite time (AUC0-∞).
Clearance rate (CL / F) | 12 hours after administration in the first and second stages
  Pharmacokinetic parameters: Clearance rate (CL / F).
apparent distribution volume (Vz / F) | 12 hours after administration in the first and second stages
  Pharmacokinetic parameters: apparent distribution volume (Vz / F).
average retention time (MRT) | 12 hours after administration in the first and second stages
  Pharmacokinetic parameters: average retention time (MRT)
Aspartate aminotransferase (AST) | after 7 days of administration in the first and 14 days of administration in second stages
  Changes in biomarkers from baseline include ALT, aspartate aminotransferase (AST).
total bilirubin (TBil) | after 7 days of administration in the first and 14 days of administration in second stages
  Changes in biomarkers from baseline include total bilirubin (TBil).
prothrombin activity (PTA) | after 7 days of administration in the first and 14 days of administration in second stages
  Changes in biomarkers from baseline include prothrombin activity (PTA).
international normalized ratio (INR) | after 7 days of administration in the first and 14 days of administration in second stages
  Changes in biomarkers from baseline include international normalized ratio (INR).
alkaline phosphatase (ALP) | after 7 days of administration in the first and 14 days of administration in second stages
  Changes in biomarkers from baseline include alkaline phosphatase (ALP)
Alpha-fetoprotein(AFP) | after 7 days of administration in the first and 14 days of administration in second stages
  Changes in biomarkers from baseline include Alpha-fetoprotein (AFP).
CK-18 M30 | after 7 days of administration in the first and 14 days of administration in second stages
  Changes in biomarkers from baseline include c aspase digested keratin 18M 30 (CK-18 M30)
caspase 3 | after 7 days of administration in the first and 14 days of administration in second stages
  Changes in biomarkers from baseline include caspase 3
caspase 1 | after 7 days of administration in the first and 14 days of administration in second stages
  Changes in biomarkers from baseline include caspase 1.
hepatocyte growth factor (HGF) | after 7 days of administration in the first and 14 days of administration in second stages
  Changes in biomarkers from baseline include hepatocyte growth factor (HGF)
the end-stage liver disease model (MELD) score | 7 days of administration in the third stage secondary outcome
  Changes of the end-stage liver disease model (MELD) score. Higher scores indicate more severe disease.
the end-stage liver disease model (MELD) score | 14 days of administration in the third stage secondary outcome
  Changes of the end-stage liver disease model (MELD) score. Higher scores indicate more severe disease.
the end-stage liver disease model (MELD) score | 28 days of administration in the third stage secondary outcome
  Changes of the end-stage liver disease model (MELD) score. Higher scores indicate more severe disease.
the end-stage liver disease model (MELD) score | 28 days of follow-up in the third stage secondary outcome
  Changes of the end-stage liver disease model (MELD) score. Higher scores indicate more severe disease.
the end-stage liver disease model (MELD) score | 90 days of follow-up in the third stage secondary outcome
  Changes of the end-stage liver disease model (MELD) score. Higher scores indicate more severe disease.
ACLF Research Consortium (AARC) score | 7 days of administration in the third stage
  Changes of ACLF Research Consortium (AARC) score. Higher scores indicate more severe disease.
ACLF Research Consortium (AARC) score | 14 days of administration in the third stage
  Changes of ACLF Research Consortium (AARC) score. Higher scores indicate more severe disease.
ACLF Research Consortium (AARC) score | 28 days of administration in the third stage
  Changes of ACLF Research Consortium (AARC) score. Higher scores indicate more severe disease.
ACLF Research Consortium (AARC) score | 28 days of follow-up in the third stage
  Changes of ACLF Research Consortium (AARC) score. Higher scores indicate more severe disease.
ACLF Research Consortium (AARC) score | 90 days of follow-up in the third stage
  Changes of ACLF Research Consortium (AARC) score. Higher scores indicate more severe disease.
Basin alanine aminotransferase (ALT) and aspartate aminotransferase (AST) | 7 days of administration in the third stage
  Changes in biomarkers compared to baseline include ALT and AST.
Basin alanine aminotransferase (ALT) and aspartate aminotransferase (AST) | 14 days of administration in the third stage
  Changes in biomarkers compared to baseline include ALT and AST.
Basin alanine aminotransferase (ALT) and aspartate aminotransferase (AST) | 28 days of administration in the third stage
  Changes in biomarkers compared to baseline include ALT and AST.
Basin alanine aminotransferase (ALT) and aspartate aminotransferase (AST) | 28 days of follow-up in the third stage
  Changes in biomarkers compared to baseline include ALT and AST.
Basin alanine aminotransferase (ALT) and aspartate aminotransferase (AST) | 90 days of follow-up in the third stage
  Changes in biomarkers compared to baseline include ALT and AST.
total bilirubin (TBil) | 7 days of administration in the third stage
  Changes in biomarkers compared to baseline include TBil.
total bilirubin (TBil) | 14 days of administration in the third stage
  Changes in biomarkers compared to baseline include TBil.
total bilirubin (TBil) | 28 days of administration in the third stage
  Changes in biomarkers compared to baseline include TBil.
total bilirubin (TBil) | 28 days of follow-up in the third stage
  Changes in biomarkers compared to baseline include TBil.
total bilirubin (TBil) | 90 days of follow-up in the third stage
  Changes in biomarkers compared to baseline include TBil.
prothrombin activity (PTA) | 7 days of administration in the third stage
  Changes in biomarkers compared to baseline include PTA.
prothrombin activity (PTA) | 14 days of administration in the third stage
  Changes in biomarkers compared to baseline include PTA.
prothrombin activity (PTA) | 28 days of administration in the third stage
  Changes in biomarkers compared to baseline include PTA.
prothrombin activity (PTA) | 28 days of follow-up in the third stage
  Changes in biomarkers compared to baseline include PTA.
prothrombin activity (PTA) | 90 days of follow-up in the third stage
  Changes in biomarkers compared to baseline include PTA.
international normalized ratio (INR) | 7 days of administration in the third stage
  Changes in biomarkers compared to baseline include international normalized ratio (INR).
international normalized ratio (INR) | 14 days of administration in the third stage
  Changes in biomarkers compared to baseline include international normalized ratio (INR).
international normalized ratio (INR) | 28 days of administration in the third stage
  Changes in biomarkers compared to baseline include international normalized ratio (INR).
international normalized ratio (INR) | 90 days of follow-up in the third stage
  Changes in biomarkers compared to baseline include international normalized ratio (INR).
alkaline phosphatase (ALP) | 7 days of administration in the third stage
  Changes in biomarkers compared to baseline include alkaline phosphatase (ALP).
alkaline phosphatase (ALP) | 14 days of administration in the third stage
  Changes in biomarkers compared to baseline include alkaline phosphatase (ALP).
alkaline phosphatase (ALP) | 28 days of administration in the third stage
  Changes in biomarkers compared to baseline include alkaline phosphatase (ALP).
alkaline phosphatase (ALP) | 28 days of follow-up in the third stage
  Changes in biomarkers compared to baseline include alkaline phosphatase (ALP).
alkaline phosphatase (ALP) | 90 days of follow-up in the third stage
  Changes in biomarkers compared to baseline include alkaline phosphatase (ALP).
Alpha-fetoprotein(AFP) | 7 days of administration in the third stage
  Changes in biomarkers compared to baseline include Alpha-fetoprotein(AFP) .
Alpha-fetoprotein(AFP) | 14 days of administration in the third stage
  Changes in biomarkers compared to baseline include Alpha-fetoprotein(AFP) .
Alpha-fetoprotein(AFP) | 28 days of administration in the third stage
  Changes in biomarkers compared to baseline include Alpha-fetoprotein(AFP) .
Alpha-fetoprotein(AFP) | 28 days of follow-up in the third stage
  Changes in biomarkers compared to baseline include Alpha-fetoprotein(AFP) .
Alpha-fetoprotein(AFP) | 90 days of follow-up in the third stage
  Changes in biomarkers compared to baseline include Alpha-fetoprotein(AFP) .
CK-18 M30 | 7 days of administration in the third stage
  Changes in biomarkers from baseline include c aspase digested keratin 18M 30 (CK-18 M30)
CK-18 M30 | 14 days of administration in the third stage
  Changes in biomarkers from baseline include c aspase digested keratin 18M 30 (CK-18 M30)
CK-18 M30 | 28 days of administration in the third stage
  Changes in biomarkers from baseline include c aspase digested keratin 18M 30 (CK-18 M30)
CK-18 M30 | 28 days of follow-up in the third stage
  Changes in biomarkers from baseline include c aspase digested keratin 18M 30 (CK-18 M30)
CK-18 M30 | 90 days of follow-up in the third stage
  Changes in biomarkers from baseline include c aspase digested keratin 18M 30 (CK-18 M30)
caspase 3 | 7 days of administration in the third stage
  Changes in biomarkers from baseline include caspase 3
caspase 3 | 14 of administration in the third stage
  Changes in biomarkers from baseline include caspase 3
caspase 3 / 7 | 28 days of administration in the third stage
  Changes in biomarkers from baseline include caspase 3
caspase 3 | 28 days of follow-up in the third stage
  Changes in biomarkers from baseline include caspase 3
caspase 3 | 90 days of follow-up in the third stage
  Changes in biomarkers from baseline include caspase 3
caspase 1 | 7 days of administration in the third stage
  Changes in biomarkers from baseline include caspase 1.
caspase 1 | 14 days of administration in the third stage
  Changes in biomarkers from baseline include caspase 1.
caspase 1 | 28 days of administration in the third stage
  Changes in biomarkers from baseline include caspase 1.
caspase 1 | 28 days of follow-up in the third stage
  Changes in biomarkers from baseline include caspase 1.
caspase 1 | 90 days of follow-up in the third stage
  Changes in biomarkers from baseline include caspase 1.
hepatocyte growth factor (HGF) | 7 days of administration in the third stage
  Changes in biomarkers from baseline include hepatocyte growth factor (HGF)
hepatocyte growth factor (HGF) | 14 days of administration in the third stage
  Changes in biomarkers from baseline include hepatocyte growth factor (HGF)
hepatocyte growth factor (HGF) | 28 days of administration in the third stage
  Changes in biomarkers from baseline include hepatocyte growth factor (HGF)
hepatocyte growth factor (HGF) | 28 days of follow-up in the third stage
  Changes in biomarkers from baseline include hepatocyte growth factor (HGF)
hepatocyte growth factor (HGF) | 90 days of follow-up in the third stage
  Changes in biomarkers from baseline include hepatocyte growth factor (HGF)
Adverse events (AE), serious adverse events (SAE) | 28 days of follow-up in the third stage.
  Adverse events (AE), serious adverse events (SAE) in the third stage at 28 days
Adverse events (AE), serious adverse events (SAE) | 90 days of follow-up in the third stage.
  Adverse events (AE), serious adverse events (SAE) in the third stage at 28 days
clinical laboratory tests ：blood routine | 28 days of follow-up ihe third stage.
  blood routine report contains the following values: RBC,WBC,NE%,LY%,HGB,PLT.
clinical laboratory tests ：blood routine | 90 days of follow-up ihe third stage.
  blood routine report contains the following values: RBC,WBC,NE%,LY%,HGB,PLT.
clinical laboratory tests ：blood biochemistry | 28 of follow-up ihe third stage.
  blood biochemistry report contains the following values: DBIL,TBIL,Urea，BUN,Cr，AST，ALT，GGT, TP, ALB, GLU,TG, TC, K,Na,CI, UA,LDH, ALP, PAB, RBP, AFP.
clinical laboratory tests ：blood biochemistry | 90 days of follow-up ihe third stage.
  blood biochemistry report contains the following values: DBIL,TBIL,Urea，BUN,Cr，AST，ALT，GGT, TP, ALB, GLU,TG, TC, K,Na,CI, UA,LDH, ALP, PAB, RBP, AFP.
clinical laboratory tests ：urine routine | 28 days of follow-up ihe third stage.
  urine routine report contains the following values: GLU,PRO,RBC,WBC.
clinical laboratory tests ：urine routine | 90 days of follow-up ihe third stage.
  urine routine report contains the following values: GLU,PRO,RBC,WBC.
clinical laboratory tests ：blood coagulation function | 28 days of follow-up ihe third stage.
  blood coagulation function report contains the following values: TT, APTT, PT, INR.
clinical laboratory tests ：blood coagulation function | 90 days of follow-up ihe third stage.
  blood coagulation function report contains the following values: TT, APTT, PT, INR.
12-lead electrocardiogram (ECG) | 28 days of follow-up ihe third stage.
  12-lead electrocardiogram (ECG) report contains the following values: HR, BP,DP,PR intervals,QRS intervals,QT intervals,QTc intervals.
12-lead electrocardiogram (ECG) | 90 days of follow-up ihe third stage.
  12-lead electrocardiogram (ECG) report contains the following values: HR, BP,DP,PR intervals,QRS intervals,QT intervals,QTc intervals.

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Beijing You 'an Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Qingyuan People's Hospital (Sixth Affiliated Hospital of Guangzhou Medical University), Qingyuan, Guangdong
  - Shiyan City Taihe Hospital, Shiyan, Hubei
  - Hunan Medical College General Hospital (formerly Huaihua City First People's Hospital), Huaihua, Hunan
  - Pingxiang Second People's Hospital, Pingxiang, Jiangxi P
  - First Hospital of Jilin University, Changchun, Jilin
  - The Affiliated Hospital of Binzhou Medical University, Binzhou, Shandong
  - Heze Municipal Hospital, Heze, Shandong
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan

IPD SHARING:
Plan to Share IPD: No